CLINICAL TRIAL: NCT05574972
Title: A Prospective, Multi-center and Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Timing Carotid Stent for Carotid Artery Stenosis（Timing Trial）
Brief Title: Timing Carotid Stent Clinical Study for the Treatment of Carotid Artery Stenosis（Timing Trial）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zenith Vascular Scitech Co., Ltd. (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTYL202201
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Carotid Artery Diseases; Carotid Artery Stenosis; Stroke; Ischemic Stroke
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Timing Carotid Stent (Experimental)
  Interventions: Device: Timing Carotid Stent
- Carotid Wallstent (Active Comparator)
  Interventions: Device: Carotid Wallstent

INTERVENTIONS:
Device: Timing Carotid Stent — all the participants in this group will be performed with Timing Carotid Stent
  Arms: Timing Carotid Stent
Device: Carotid Wallstent — all the participants in this group will be performed with Carotid Wallstent
  Arms: Carotid Wallstent

SUMMARY:
Evaluate the safety and efficacy of the Timing Carotid Stent for the treatment of carotid artery stenosis in patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, concurrent controlled, multi-center study. Patients with carotid artery stenosis will be assigned to either the Timing Carotid Stent or Carotid Wallstent. Each treated patient will be followed and assessed for 12 months after randomization. The hypothesis to be tested is that the safety and effectiveness of the Timing Carotid Stent is not inferior to the Carotid Wallstent.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years;
2. Patient is either symptomatic with carotid stenosis ≥50% OR asymptomatic with carotid stenosis ≥70% ;
3. Target lesion 3.5- 5.5 mm;
4. Signed informed consent.

Exclusion Criteria:

1. Target lesion is not caused by atherosclerotic disease；
2. Target lesion is located at the opening of the common carotid artery；
3. Patient has severe lesion calcification that may restrict the full deployment of the carotid
4. Patient has a total occlusion of the target carotid arteries
5. Patient has a large number of acute or subacute thrombi and arteriovenous malformations near the target lesion
6. Patient has a severe stenosis or occlusion in series with target lesions
7. Patient has known severe carotid stenosis contralateral to the target lesion
8. Patient need angioplasty in other parts (including intracranial and extracranial) at the same time or within 30 days after procedure
9. Patient has a symptomatic severe stenosis of other blood vessels (including intracranial and extracranial) except carotid artery
10. Patient is experiencing (or has experienced) an evolving, acute, or recent disabling stroke or intracranial hemorrhage
11. Patient has a massive stroke or myocardial infarction
12. Patient has a intracranial aneurysm
13. Patient has a coagulation dysfunction or abnormal bleeding, or contraindications to heparin and antiplatelet drugs
14. Patient has known sensitivity to contrast agent
15. Patient has a platelet < 90 × 109 / L, severe liver and kidney injury, and severe dysfunction of important organs such as heart, lung, liver and kidney
16. Patient has a uncontrollable severe hyperemia
17. Patient has a bradycardia
18. mRS≥3
19. Patient has life expectancy of less than one year
20. Patient is currently enrolled in another investigational study protocol
21. Females who are pregnant or in lactation
22. Other conditions not suitable for inclusion judged by the researcher -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Major Adverse Events (MAE) at 30 days | 30 days
  MAE defined as any death, stroke, or myocardial infarction through 30 days post-index procedure

SECONDARY OUTCOMES:
Number of Participants Who Achieved Stent Technical Success | Procedural
  Stent Technical Success defined as successful implantation of a Carotid Stent
Number of Participants Who Achieved Procedure Success | Procedural
  Number of Participants Who Achieved Procedure Success
Target Lesion Revascularization | 30 days
  Any clinically driven revascularization procedure that is performed to increase the luminal diameter inside or within 5 mm of the previously treated lesion
In-Stent Restenosis | 1 year
  ≥50% diameter stenosis within the stented lesion or within 5 mm proximal or distal to the stent at follow-up evaluation
Ipsilateral ischemic stroke | 1 year
  Any ipsilateral ischemic stroke through 1 year post-index procedure
mRS score change | 1 year
  mRS score change through 1 year post-index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No